CLINICAL TRIAL: NCT06304376
Title: Evaluation of Shell Technique for Reconstruction of Alveolar Cleft: Retrospective Study
Brief Title: Evaluation of Shell Technique in Secondary Alveolar Cleft Grafting
Acronym: Alveolar cleft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Khalid Tarek Mohamed Karkar, Priniciple investigator, Ministry of Health, Kuwait
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS/FSDC002
Record Dates: First submitted 2024-03-01; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Alveolar Cleft; Alveolar Ridge Cleft
Keywords: alveolar ridge cleft; Khoury shell technique; 3D alveolar ridge reconstruction; anterior iliac crest bone graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other): This study group contains of patient who had alveolar cleft, indicated for late secondary alveolar grafting
  Interventions: Procedure: Alveolar ridge grafting

INTERVENTIONS:
Procedure: Alveolar ridge grafting — Alveolar ridge grafting was carried out using anterior iliac crest bone graft. Khoury shell technique was the method of ridge reconstruction via a cortical bone shell was fixed away from alveolar ridge using two micro-screws and the gap created was filled by cancellous bone

SUMMARY:
This study aims to evaluate the sufficiency of Khoury shell technique for reconstruction of alveolar cleft. Khoury technique was carried out using cortical bone shell fixed away from alveolar bone using two micro-screws, which was harvested from anterior iliac bone crest. The gap between the shell cortical bone and the native alveolar bone was filled by cancellous bone which was harvested from anterior iliac crest bone. The whole graft was covered by collagen membrane. The volumetric bone gain of the defect was determined via CBCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with alveolar ridge cleft
2. Males and females 7-14 years of age.
3. Patients with adequate oral hygiene.
4. Compliance with all requirements in the study and signing the informed consent.

Exclusion Criteria:

1. Patients with diseases of the immune system or any medical condition that may influence the outcome (uncontrolled diabetes, Glycated hemoglobin- HbA1c ≥ 7%).
2. Patients with systemic disease affecting bone healing.
3. Patients who are chronic users of medications known to affect the periodontal status (calcium antagonists, anti-convulsives, immunosuppressives, anti-inflammatory medications).
4. Patients with history of intravenous and/or oral bisphosphonate use.
5. Pathologic lesions or acute infection in the area of defect.
6. Patients with poor oral hygiene that are not amenable to motivation and improvement.

8. Vulnerable patients.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Volumetric bone gain | 4 months
  bone volumetric gain and changes measured by CBCT analysis

SECONDARY OUTCOMES:
Eruption of the tooth in the cleft | 6-9 months
  Eruption of the tooth assessed clinically and radiographically

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Farwaniya Hospital, Al Farwānīyah, Kuwait

IPD SHARING:
Plan to Share IPD: No